CLINICAL TRIAL: NCT03083639
Title: A Phase 1, Randomized, Open-label, 2-way Cross-over Study to Evaluate the Bioequivalence Between a Single Oral Dose of Esomeprazole 40 mg Capsules and Esomeprazole 40 mg Tablets in Healthy Subjects
Brief Title: A Study to Evaluate the Bioequivalence of Single Oral Dose of Esomeprazole Capsule and Tablet Formulation in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Esomeprazole-1001; U1111-1189-8028 (Other: WHO); 03083639 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Healthy Participants
Keywords: Drug Therapy
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esomeprazole 40 mg Capsule + Esomeprazole 40 mg Tablet (Experimental): Esomeprazole 40 mg, capsule, orally, once on Day 1 of Intervention Period 1, followed by 6 days of washout period, followed by esomeprazole 40 mg tablet, orally, once on Day 1 of Intervention Period 2.
  Interventions: Drug: Esomeprazole Capsule; Drug: Esomeprazole Tablet
- Esomeprazole 40 mg Tablet + Esomeprazole 40 mg Capsule (Experimental): Esomeprazole 40 mg, tablet, orally, once on Day 1 of Intervention Period 1, followed by 6 days of washout period, followed by esomeprazole 40 mg capsule, orally, once on Day 1 of Intervention Period 2.
  Interventions: Drug: Esomeprazole Capsule; Drug: Esomeprazole Tablet

INTERVENTIONS:
Drug: Esomeprazole Capsule — Esomeprazole Capsule
  Other Names: Nexium
Drug: Esomeprazole Tablet — Esomeprazole Tablet
  Other Names: Nexium

SUMMARY:
The purpose of this study is to determine the bioequivalence of esomeprazole 40 milligram (mg) tablets and capsules.

DETAILED DESCRIPTION:
The drug being tested in this study is called esomeprazole. Esomeprazole is being tested in healthy participants in order to evaluate the bioequivalence between a single oral dose of esomeprazole tablet and capsule. The study will enroll 52 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment sequences:

* Esomeprazole 40 mg capsule + Esomeprazole 40 mg tablet
* Esomeprazole 40 mg tablet + Esomeprazole 40 mg capsule

All participants will be asked to take one capsule or tablet on Day 1 of each Intervention Period based on the treatment sequence to which the participant has been assigned.

This single center trial will be conducted in the United States. The overall duration to participate in this study is 36 days. Participants will visit the clinic on Day -1 and remained confined until Day 1 of Intervention Period 1 and 2. A washout period of minimum 6 days will be maintained between the dose in each Intervention Period.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult male or female participant.
2. Is aged 18 to 55 years, inclusive, at the time of informed consent and first study medication dose.
3. Weighs at least 50 kilogram (kg) and has a body mass index (BMI) from 18.5 to 30 kilogram per square meter (kg/m^2), inclusive at Screening and Day -1.

Exclusion Criteria:

1. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results. It is the responsibility of the investigator to assess the clinical significance; however, consultation with the Takeda Medical Monitor may be warranted.
2. Has a history of significant gastro intestinal (GI) disorders manifested with persistent, chronic or intermittent nausea, vomiting, diarrhea, or has a current or recent (within 6 months) GI disease that would influence the absorption of drugs (example, a history of malabsorption, severe esophageal reflux, peptic ulcer disease or erosive esophagitis), or any gastrointestinal-related surgical intervention..
3. Has a known hypersensitivity to any component of the formulation of esomeprazole capsules or tablets or compounds with the same mechanism of action (dexlansoprazole, lansoprazole, omeprazole, rabeprazole, pantoprazole), or related compounds.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-05-13 (Actual); Study Completion 2017-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Pharmaceutical Research Associates, Inc., Lenexa, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 27 March 2017 to 13 May 2017.
Pre-assignment Details: Healthy participants were enrolled in this 2-way crossover study and randomized in 1 of the 2 treatment sequences to receive esomeprazole 40 milligram (mg) capsule (Regimen A) or esomeprazole 40 mg tablet (Regimen B) under fasted conditions.
Groups:
- Regimen A + Regimen B: Esomeprazole 40 mg, capsule, orally, once under fasted conditions on Day 1 of Intervention Period 1, followed by at least 6 days of washout period, further followed by esomeprazole 40 mg, tablet, orally, once under fasted conditions on Day 1 of Intervention Period 2.
- Regimen B + Regimen A: Esomeprazole 40 mg, tablet, orally, once under fasted conditions on Day 1 of Intervention Period 1, followed by at least 6 days of washout period, further followed by esomeprazole 40 mg, capsule, orally, once under fasted conditions on Day 1 of Intervention Period 2.
Period: Intervention Period 1 (1 Day)
Arm/Group | Regimen A + Regimen B | Regimen B + Regimen A
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0
Period: Washout Period (at Least 6 Days)
Arm/Group | Regimen A + Regimen B | Regimen B + Regimen A
Started | 26 | 26
Completed | 25 | 25
Not Completed | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Intervention Period 2 (1 Day)
Arm/Group | Regimen A + Regimen B | Regimen B + Regimen A
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A + Regimen B | Regimen B + Regimen A | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  years | 32.4 (9.64) | 33.3 (7.83) | 32.8 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    Female | 9 | 11 | 20
    Male | 17 | 15 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 8 | 11 | 19
    White | 18 | 13 | 31
    More than one race | 0 | 2 | 2
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    United States | 26 | 26 | 52
Weight [Mean (Standard Deviation); unit: kilogram] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  kilogram | 73.3 (12.83) | 75.3 (13.37) | 74.3 (13.01)
Height [Mean (Standard Deviation); unit: centimeter] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  centimeter | 173.4 (10.36) | 170.7 (10.95) | 172.0 (10.65)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  kilogram per square meter (kg/m^2) | 24.3 (2.77) | 25.7 (2.89) | 25.0 (2.89)
Smoking Status [Count of Participants; unit: Participants] — Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
  Participants
    Never smoked | 18 | 24 | 42
    Ex-smoker | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Esomeprazole
Time Frame: Day 1 pre-dose and at multiple time points (up to 10 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration of study drug. The PK set where data at specified timepoints was available for all participants who received at least one dose of Regimen A and Regimen B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Regimen A: Esomeprazole 40 mg, capsule, orally, once under fasted conditions on Day 1 of either Intervention Period 1 or Intervention Period 2.
- Regimen B: Esomeprazole 40 mg, tablet, orally, once under fasted conditions on Day 1 of either Intervention Period 1 or Intervention Period 2.
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 51 | 49
hour*nanogram per milliliter (h*ng/mL) | 1908.0 (66.0) | 1922.2 (57.9)
Statistical Analysis 1: Comparison: Regimen A vs Regimen B; Test type: Equivalence — The bioequivalence between esomeprazole capsules (Regimen A) and esomeprazole tablets (Regimen B) was assessed for the natural logarithms of AUC∞ using analysis of variance (ANOVA) models. The models included regimen, period, and sequence as fixed effects and participant nested within sequence as a random effect. Within ANOVA framework, point estimates and their 90 percent (%) confidence intervals (CIs) for the ratio of AUC central values between esomeprazole capsules and tablets are presented; Point estimate = 1.018, 90% CI 2-sided [0.969 to 1.070]

2. Primary Outcome: AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t for Esomeprazole
Time Frame: Day 1 pre-dose and at multiple time points (up to 10 hours) post-dose
Population: The PK set included all participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration of study drug. The PK set where data at specified timepoints was available for all participants who received at least one dose of Regimen A and Regimen B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 51 | 51
h*ng/mL | 1884.6 (64.3) | 1882.6 (57.5)
Statistical Analysis 1: Comparison: Regimen A vs Regimen B; Test type: Equivalence — The bioequivalence between esomeprazole capsules (Regimen A) and esomeprazole tablets (Regimen B) was assessed for the natural logarithms of AUCt using ANOVA models. The models included regimen, period, and sequence as fixed effects and participant nested within sequence as a random effect. Within ANOVA framework, point estimates and their 90% CIs for the ratio of AUC central values between esomeprazole capsules and tablets are presented; Point estimate = 0.993, 90% CI 2-sided [0.939 to 1.050]

3. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Esomeprazole
Time Frame: Day 1 pre-dose and at multiple time points (up to 10 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 51 | 51
nanogram per milliliter (ng/mL) | 933.29 (44.5) | 872.38 (43.5)
Statistical Analysis 1: Comparison: Regimen A vs Regimen B; Test type: Equivalence — The bioequivalence between esomeprazole capsules (Regimen A) and esomeprazole tablets (Regimen B) was assessed for the natural logarithms of Cmax using ANOVA models. The models included regimen, period, and sequence as fixed effects and participant nested within sequence as a random effect. Within ANOVA framework, point estimates and their 90% CIs for the ratio of Cmax central values between esomeprazole capsules and tablets are presented; Point estimate = 0.942, 90% CI 2-sided [0.880 to 1.009]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. The safety set where data was available for all participants who received at least one dose of Regimen A and Regimen B.
Arm/Group | Regimen A | Regimen B
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 4/51 | 3/51
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A (N=51) | Regimen B (N=51)
Headache (Nervous system disorders) | 3 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03083639/SAP_000.pdf
  • Study Protocol (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT03083639/Prot_001.pdf